CLINICAL TRIAL: NCT04469803
Title: The Impact of Napping During Night Shifts on Indicators of Cardiovascular Health Among EMS Clinicians
Brief Title: Impact of Intra-Shift Napping on EMS Cardiovascular Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: ZOLL Foundation (Unknown)
Responsible Party: Principal Investigator, Leonard Weiss, Assistant Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: STUDY19120222
Record Dates: First submitted 2020-07-09; First posted 2020-07-14 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Blood Pressure; Heart Rate Variability

STUDY DESIGN:
Intervention Model Description: Randomized crossover study design
Masking Description: No masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- No nap, brief nap, then longer nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with no nap first, undergo a 1-week minimum washout, then complete the protocol again with a brief nap, then undergo a minimum 1-week washout, then return to complete the protocol again with a longer nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping
- No nap, longer nap, then brief nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with no nap first, undergo a 1-week minimum washout, then complete the protocol again with a longer nap, then undergo a minimum 1-week washout, then return to complete the protocol again with a brief nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping
- Brief nap, no nap, then longer nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with brief nap first, undergo a 1-week minimum washout, then complete the protocol again with no nap, then undergo a minimum 1-week washout, then return to complete the protocol again with a longer nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping
- Brief nap, longer nap, then no nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with brief nap first, undergo a 1-week minimum washout, then complete the protocol again with longer nap, then undergo a minimum 1-week washout, then return to complete the protocol again with no nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping
- Longer nap, brief nap, then no nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with a longer nap first, undergo a 1-week minimum washout, then complete the protocol again with a brief nap, then undergo a minimum 1-week washout, then return to complete the protocol again with no nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping
- Longer nap, no nap, then brief nap (Experimental): Participants will be monitored for 72 total hours, including a 12-hour simulated night shift. At baseline (consent), participants randomized to crossover study design with three study arms (No nap, brief nap, longer nap). In this sequence, participants will perform the 12-hour night shift with a longer nap first, undergo a 1-week minimum washout, then complete the protocol again with no nap, then undergo a minimum 1-week washout, then return to complete the protocol again with a brief nap opportunity.
  Interventions: Behavioral: Intra-Shift Napping

INTERVENTIONS:
Behavioral: Intra-Shift Napping — The Brief Nap opportunity will allow for a 30-minute nap between the hours of 0200 and 0400 during the 12-hour simulated night shift. The Longer Nap opportunity will allow for a 2-hour nap between the hours of 0200 and 0400 during the 12-hour simulated night shift.

SUMMARY:
Cardiovascular disease (CVD) exerts a significant health burden among shift workers, including police, firefighters, and emergency medical services (EMS). The unique occupational demands inherent to these professions--sleep loss, circadian misalignment, high stress, and sustained hyper-vigilance--confer increased risk for both on and off-duty cardiovascular events. Mitigating cardiovascular risks in these professions requires that we first identify robust markers and potential mechanisms of risk. Previous work suggest shift work has a negative impact on blood pressure (BP) and heart rate variability (HRV). Blunted BP dipping at night and during sleep, and reduced HRV are powerful markers of increased CVD risk. Both are linked to preclinical indicators of cardiac damage, such as presence of coronary artery calcium, left atrial enlargement, and cardiovascular-related mortality. This study will use an experimental crossover study design with three intervention conditions to test the impact of a 30 minute brief nap and a 2-hour longer nap versus no nap on BP and HRV. Outcomes of interest include blunted dipping of BP during nighttime hours and during sleep and HRV.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) exerts a significant health burden among shift workers, including police, firefighters, and emergency medical services (EMS). The unique occupational demands inherent to these professions--sleep loss, circadian misalignment, high stress, and sustained hyper-vigilance--confer increased risk for both on and off-duty cardiovascular events. Mitigating cardiovascular risks in these professions requires that we first identify robust markers and potential mechanisms of risk. Previous work suggest shift work has a negative impact on blood pressure (BP) and heart rate variability (HRV). Blunted BP dipping at night and during sleep, and reduced HRV are powerful markers of increased CVD risk. Both are linked to preclinical indicators of cardiac damage, such as presence of coronary artery calcium, left atrial enlargement, and cardiovascular-related mortality.

Critical questions remain:

Are BP dipping and HRV impacted by napping during night shift work? Compared to those who do not nap, does napping during night shifts help BP and HRV to normalize quicker in the hours immediately post night shift work? What is the impact of brief naps (e.g., 30 minutes) versus longer naps (e.g., 2 hours)?

This study will use a randomized crossover experimental design of EMS workers and be based in the laboratory environment. Participants will complete three intervention conditions. All study arms will involve a 12-hour simulated night shift. The intervention of interest is napping (no nap vs. a 30 minute nap vs. a two-hour nap) in a randomized crossover study design. The primary outcome of interest is BP dipping (>10% drop) and Heart Rate Variability (HRV) measured as the standard deviation of inter-beat intervals of the sinus beats in milliseconds (SDNN). All outcomes will be measured serially before the simulation, during simulated night shifts, during the intra-shift napping period, and during recovery.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 years or older;
2. current / active certification as an EMS clinician at the EMT-Basic, Advanced, Paramedic, Flight Paramedic, or Flight Nurse level, or healthcare shift worker;
3. has not ever been diagnosed with any of the following: hypertension, cardiovascular disease, myocardial infarction, stroke/TIA, chronic kidney disease, adrenal disease, thyroid disease, rheumatologic disease, hematologic disease, cancer of any type, dementia/memory loss, organ transplantation; insomnia or other major sleep problem; sleep apnea or other diagnosis that is related to problems with breathing or the airway; and
4. is not currently pregnant.

Exclusion Criteria:

1. 17 years of age or younger;
2. not an EMS clinician or inactive as an EMS clinician or not a healthcare shift worker;
3. has ever been diagnosed with hypertension, cardiovascular disease, myocardial infarction, stroke/TIA, chronic kidney disease, adrenal disease, thyroid disease, rheumatologic disease, hematologic disease, cancer of any type, dementia/memory loss, organ transplantation; insomnia or other major sleep problem; sleep apnea or other diagnosis that is related to problems with breathing or the airway;
4. is currently pregnant;
5. is unwilling to wear multiple monitoring devices (e.g., automated blood pressure monitoring device, holter monitor for HRV measurement, wrist actigraphy) for the duration of the study protocol.
6. is unwilling to refrain from caffeine during the study protocol; or
7. is unwilling to adhere to sleep / wake times outlined in the study protocol.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-10-02 (Actual); Study Completion 2022-10-02 (Actual)

PRIMARY OUTCOMES:
Number of participants with blunted dipping of blood pressure via the sleep based method | Blood pressure will be monitored with automated devices at 1-hour intervals over 72 total hours
  Blood pressure is created by the heart muscle contractions and is measured using two numbers: The Systolic Blood Pressure (SBP) and the Diastolic Blood Pressure (DBP). Normal patterns in BP include elevations in SBP and DBP during the daylight and waking hours followed by a drop (dip) during nighttime hours and during sleep. A dip of 10% to 20% during nighttime or sleep is considered normal, whereas a dip <10% is defined as blunted BP dipping. Blunted BP dipping will be quantified as: [(mean BP during waking hours - mean BP during sleep) / mean BP during waking hours] X 100 - the "sleep-based method."
Number of participants with blunted dipping of blood pressure via the wide fixed time method | Blood pressure will be monitored with automated devices at 1-hour intervals over 72 total hours
  Blood pressure is created by the heart muscle contractions and is measured using two numbers: The Systolic Blood Pressure (SBP) and the Diastolic Blood Pressure (DBP). Normal patterns in BP include elevations in SBP and DBP during the daylight and waking hours followed by a drop (dip) during nighttime hours and during sleep. A dip of 10% to 20% during nighttime or sleep is considered normal, whereas a dip <10% is defined as blunted BP dipping. Blunted BP dipping during nighttime hours (2300 to 0659 hours) vs. daytime hours (0700 to 2259 hours) will be quantified as: [(mean daytime BP - mean nighttime BP) / mean daytime hours BP] X 100 - the "wide-fixed time method."
The number of participants with unhealthy Heart Rate Variability (HRV) measured via the standard deviation of the inter-beat intervals of normal sinus beats (SDNN) | HRV will be monitored with a holter monitor continuously over 72 total hours
  A healthy heart oscillates and beat-to-beat fluctuations are variable. Greater variability in heart rate is associated with better health, the capacity to respond and cope, and better performance. The Heart Rate Variability (HRV) measure standard deviation of the inter-beat intervals of normal sinus beats (SDNN) is considered standard and is calculated in milliseconds (ms) over short-term (e.g., 60 seconds) and long-term intervals (24 hours). Values of SDNN <50ms are considered unhealthy for medical risk stratification.

CONTACTS AND LOCATIONS:
Overall Officials: Leonard Weiss, MD, Principal Investigator — University of Pittsburgh; P. Daniel Patterson, PhD, Study Director — University of Pittsburgh
Locations (1):
- University of Pittsburgh, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will work with the ZOLL Foundation and share de-identified research data if requested and if approved by the University of Pittsburgh. The study team will develop a process to receive requests from outside the study team for de-identified datasets.
Supporting Information: Study Protocol, SAP
Time Frame: One year after the main results are reported in peer-reviewed manuscripts.
Access Criteria: The study team will develop a process to receive requests from outside the study team for de-identified datasets.

REFERENCES:
- [Background] Patterson PD, Weiss LS, Weaver MD, Salcido DD, Opitz SE, Okerman TS, Smida TT, Martin SE, Guyette FX, Martin-Gill C, Callaway CW. Napping on the night shift and its impact on blood pressure and heart rate variability among emergency medical services workers: study protocol for a randomized crossover trial. Trials. 2021 Mar 16;22(1):212. doi: 10.1186/s13063-021-05161-4. PMID 33726840
- [Derived] Patterson PD, Okerman TS, Roach DGL, Hilditch CJ, Weaver MD, Patterson CG, Sheffield MA, Di Salvatore JS, Bernstein H, Georges G, Andreozzi A, Willson CM, Jain D, Martin SE, Weiss LS. Are Short Duration Naps Better than Long Duration Naps for Mitigating Sleep Inertia? Brief Report of a Randomized Crossover Trial of Simulated Night Shift Work. Prehosp Emerg Care. 2023;27(6):807-814. doi: 10.1080/10903127.2023.2227696. Epub 2023 Jul 17. PMID 37347968
- [Derived] Patterson PD, Okerman TS, Roach DGL, Weaver MD, Patterson CG, Martin SE, Okwiya N, Nong L, Eyiba C, Huff JR, Ruzicka A, Ruggieri J, McIlvaine Q, Weiss LS. Effect of Short versus Long Duration Naps on Blood Pressure during Simulated Night Shift Work: A Randomized Crossover Trial. Prehosp Emerg Care. 2023;27(6):815-824. doi: 10.1080/10903127.2023.2227891. Epub 2023 Jul 17. PMID 37347964